CLINICAL TRIAL: NCT05477992
Title: Haemorrhage Risk Reduction Using Endovascular Embolisation in Place of Vessel Ligation for Patients Undergoing Transoral Robotic Surgery (HELPR)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCR5262
Record Dates: First submitted 2022-07-20; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Non-randomised interventional feasibility study at a single institution
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovascular embolisation (Experimental): Embolisation is an effective measure to reduce intraoperative bleeding for vascular tumours of the head and neck. It is often carried out from 24 to 72 hours prior to the surgical resection to allow time for maximal thrombosis of the occluded vessels and prevent recanalisation of the occluded arteries or formation of collateral arterial channels. Data will be collected for primary and secondary outcome measures
  Interventions: Procedure: Endovascular embolization

INTERVENTIONS:
Procedure: Endovascular embolization — Embolisation is an effective measure to reduce intraoperative bleeding for vascular tumours of the head and neck. It is often carried out from 24 to 72 hours prior to the surgical resection to allow time for maximal thrombosis of the occluded vessels and prevent recanalisation of the occluded arteries or formation of collateral arterial channels.

SUMMARY:
Transoral robotic surgery (TORS )has been shown to offer excellent oncological and functional outcomes for treating cancer at multiple subsites of the head and neck. Post operative haemorrhage (3.1% to 13.1%) is the most common complication of this procedure and can lead to airway compromise. Ligation of individual feeding vessels in the neck can limit risk of severe bleed and is usually done when concomitant neck dissection is carried out with TORS. In salvage TORS, in the absence of any nodal disease of the neck, the neck is explored, nevertheless, for the sole purpose of tying the vessel. Endovascular embolisation is a minimally invasive, safe and effective procedure; known for treating refractory epistaxis and for reducing intra-operative bleeding for benign vascular head and neck tumour. The investigators propose that superselective endovascular embolisation to occlude feeding blood vessels prior to TORS in patients who do not require neck dissection is a feasible, safe and acceptable intervention; and therefore a plausible alternative conventional open neck vessel ligation.

DETAILED DESCRIPTION:
The incidence of squamous cell carcinoma of oropharynx has increased at an alarming rate attributed to human papillomavirus (HPV).The prognosis of patients with HPV-associated oropharyngeal cancer is significantly improved, and as such, consideration of functional outcomes has become increasingly important. Transoral robotic surgery (TORS) has been shown to offer excellent oncological outcomes and low incidence of positive margins with promising functional outcome at multiple subsites of the head and neck. Like many oropharyngeal surgeries, bleeding is the most common complication after TORS. Postoperative oropharyngeal haemorrhage, particularly when severe, can lead to airway compromise, aspiration, asphyxiation, and cardiopulmonary arrest. Its incidence has been variable in literature, with rates ranging from 3.1% to 13.1%. It is an area of current interest because of the increasing adoption of TORS and the active recruitment to current multi-centre randomized controlled trials, such as ECOG 3311 (NCT01898494) and PATHOS. Ligation of the individual feeding vessels from the external carotid artery (e.g. ascending pharyngeal, lingual and facial branches) has shown to limit the risk of postoperative haemorrhage and is highly recommended. This is usually done when concomitant neck dissection is carried out with transoral resection. However, in the absence of any nodal disease, for instance in salvage TORS for recurrent oropharyngeal cancer, the neck is surgically explored for the sole purpose of tying the vessel. This is particularly more difficult surgically and carries a higher risk of failure in patients who had exposure to prior radiation where healing can be dramatically delayed. Embolisation, first described in 1974, is now a well-recognised treatment for refractory epistaxis and an effective measure to reduce intraoperative bleeding for vascular tumours of the head and neck. The latter is often carried out from 24 to 72 hours prior to the surgical resection to allow time for maximal thrombosis of the occluded vessels and prevent recanalization of the occluded arteries or formation of collateral arterial channels. This procedure has been proven to be minimally invasive, safe and effective in controlling haemorrhage even in cases of acute carotid blowout syndrome. The targeted vessels for embolisation are also branches of the external carotid artery, of similar calibre and size to the feeding vessels which are ligated in TORS. Although endovascular embolisation of branches of external carotid artery has not been carried out for the purpose of TORS in the past, it has been highly successful in controlling of bleeding in the case of benign vascular tumours of head and head. The investigators propose that this standard endovascular embolisation can also be applied to patient undergoing TORS who do not require neck dissection. The investigators believe that this is a feasible, safe and acceptable intervention and a plausible alternative to conventional open neck vessel ligation.

ELIGIBILITY:
For Main Study:

Inclusion Criteria

* Residual, recurrent or new primary oropharyngeal, laryngeal or hypopharyngeal cancer, in a previously irradiated field.
* Listed for TORS resection
* Who would normally be indicated for concurrent ligation of branches of their external carotid artery for peri-operative haemorrhage control

Exclusion Criteria

* Patients requiring concurrent ipsilateral neck surgery alongside their TORS resection, who would be more suited to undergo surgical vessel ligation.
* Patients known to have undergone previous ligation or embolisation of the ipsilateral external carotid artery or the relevant feeding branches.
* Females who are pregnant
* Females of childbearing potential should only be included after a confirmed menstrual period and a negative highly sensitive urine or serum pregnancy test
* Females must not be breastfeeding.

For Retrospective Sub-Study

Inclusion Criteria

* Residual, recurrent or new primary oropharyngeal, laryngeal or hypopharyngeal cancer, in a previously irradiated field
* Who underwent TORS resection to manage this disease
* Who had concurrent neck surgery for surgical ligation of branches of their external carotid artery for peri-operative haemorrhage control

Exclusion Criteria

- Patients known to have undergone previous ligation or embolisation of the ipsilateral external carotid artery or the relevant feeding branches.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of embolisation procedure | Day 1 post the embolisation procedure
  Measure by the calculating the proportion of successful completion of embolisation procedure out of the total number of patients eligible for the embolisation procedure.
Feasibility of open neck vessel ligation | Day 1 post open neck vessel ligation
  Measure by the calculating the proportion of successful completion of open neck vessel ligation procedure out of the total number of patients who undergo this procedure.

SECONDARY OUTCOMES:
Safety of embolisation procedure | Day 30 post embolisation procedure
  Measured by calculating the proportion of major or minor adverse event sites out of all patients who undergo embolisation
Efficacy of embolisation procedure | Day 30 post embolisation procedure
  Measured by calculating the proportion of post-operative bleeding from the primary site in all patients who undergo embolisation
Acceptability of embolisation procedure | After day 30 post procedure, at the time of focus group discussion
  Qualitative methods only, therefore no quantitative endpoint
Safety of open neck vessel ligation | Day 30 post open neck vessel ligation
  Measured by calculating the proportion of major or minor adverse event sites out of all patients who undergo open neck vessel ligation
Efficacy of open neck vessel ligation | Day 30 post open neck vessel ligation
  Measured by calculating the proportion of major or minor adverse event sites out of all patients who undergo open neck vessel ligation

CONTACTS AND LOCATIONS:
Overall Officials: Vinidh Paleri, Principal Investigator — Royal Marsden NHS Foundation Trust

REFERENCES:
- [Background] Pytynia KB, Dahlstrom KR, Sturgis EM. Epidemiology of HPV-associated oropharyngeal cancer. Oral Oncol. 2014 May;50(5):380-6. doi: 10.1016/j.oraloncology.2013.12.019. Epub 2014 Jan 22. PMID 24461628
- [Background] D'Souza G, Kreimer AR, Viscidi R, Pawlita M, Fakhry C, Koch WM, Westra WH, Gillison ML. Case-control study of human papillomavirus and oropharyngeal cancer. N Engl J Med. 2007 May 10;356(19):1944-56. doi: 10.1056/NEJMoa065497. PMID 17494927
- [Background] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Background] de Almeida JR, Byrd JK, Wu R, Stucken CL, Duvvuri U, Goldstein DP, Miles BA, Teng MS, Gupta V, Genden EM. A systematic review of transoral robotic surgery and radiotherapy for early oropharynx cancer: a systematic review. Laryngoscope. 2014 Sep;124(9):2096-102. doi: 10.1002/lary.24712. Epub 2014 May 27. PMID 24729006
- [Background] Kelly K, Johnson-Obaseki S, Lumingu J, Corsten M. Oncologic, functional and surgical outcomes of primary Transoral Robotic Surgery for early squamous cell cancer of the oropharynx: a systematic review. Oral Oncol. 2014 Aug;50(8):696-703. doi: 10.1016/j.oraloncology.2014.04.005. Epub 2014 Jun 7. PMID 24917389
- [Background] Hutcheson KA, Holsinger FC, Kupferman ME, Lewin JS. Functional outcomes after TORS for oropharyngeal cancer: a systematic review. Eur Arch Otorhinolaryngol. 2015 Feb;272(2):463-71. doi: 10.1007/s00405-014-2985-7. Epub 2014 Mar 19. PMID 24643851
- [Background] Weinstein GS, O'Malley BW Jr, Magnuson JS, Carroll WR, Olsen KD, Daio L, Moore EJ, Holsinger FC. Transoral robotic surgery: a multicenter study to assess feasibility, safety, and surgical margins. Laryngoscope. 2012 Aug;122(8):1701-7. doi: 10.1002/lary.23294. Epub 2012 Jul 2. PMID 22752997
- [Background] Chia SH, Gross ND, Richmon JD. Surgeon experience and complications with Transoral Robotic Surgery (TORS). Otolaryngol Head Neck Surg. 2013 Dec;149(6):885-92. doi: 10.1177/0194599813503446. Epub 2013 Sep 6. PMID 24013139
- [Background] Pollei TR, Hinni ML, Moore EJ, Hayden RE, Olsen KD, Casler JD, Walter LC. Analysis of postoperative bleeding and risk factors in transoral surgery of the oropharynx. JAMA Otolaryngol Head Neck Surg. 2013 Nov;139(11):1212-8. doi: 10.1001/jamaoto.2013.5097. PMID 24113922
- [Background] Laccourreye O, Malinvaud D, Garcia D, Menard M, Hans S, Cauchois R, Bonfils P. Postoperative hemorrhage after transoral oropharyngectomy for cancer of the lateral oropharynx. Ann Otol Rhinol Laryngol. 2015 May;124(5):361-7. doi: 10.1177/0003489414558109. Epub 2014 Nov 10. PMID 25385839
- [Background] Asher SA, White HN, Kejner AE, Rosenthal EL, Carroll WR, Magnuson JS. Hemorrhage after transoral robotic-assisted surgery. Otolaryngol Head Neck Surg. 2013 Jul;149(1):112-7. doi: 10.1177/0194599813486254. Epub 2013 Apr 12. PMID 23585156
- [Background] Lorincz BB, Mockelmann N, Busch CJ, Knecht R. Functional outcomes, feasibility, and safety of resection of transoral robotic surgery: single-institution series of 35 consecutive cases of transoral robotic surgery for oropharyngeal squamous cell carcinoma. Head Neck. 2015 Nov;37(11):1618-24. doi: 10.1002/hed.23809. Epub 2014 Aug 28. PMID 24955923
- [Background] Mandal R, Duvvuri U, Ferris RL, Kaffenberger TM, Choby GW, Kim S. Analysis of post-transoral robotic-assisted surgery hemorrhage: Frequency, outcomes, and prevention. Head Neck. 2016 Apr;38 Suppl 1:E776-82. doi: 10.1002/hed.24101. Epub 2015 Jul 15. PMID 25916790
- [Background] ECOG-ACRIN E3311: Phase II Randomized Trial of Transoral Surgical Resection Followed by Low-dose or Standard-dose IMRT in Resectable p16+ Locally Advanced Oropharynx Cancer [Internet]. [cited 2019 Nov 24];Available from: https://www.cityofhope.org/clinical-trial/ecog-acrin-e3311:-phase-ii-randomized-trial-of-transoral-sur
- [Background] Owadally W, Hurt C, Timmins H, Parsons E, Townsend S, Patterson J, Hutcheson K, Powell N, Beasley M, Palaniappan N, Robinson M, Jones TM, Evans M. PATHOS: a phase II/III trial of risk-stratified, reduced intensity adjuvant treatment in patients undergoing transoral surgery for Human papillomavirus (HPV) positive oropharyngeal cancer. BMC Cancer. 2015 Aug 27;15:602. doi: 10.1186/s12885-015-1598-x. PMID 26311526
- [Background] Kubik M, Mandal R, Albergotti W, Duvvuri U, Ferris RL, Kim S. Effect of transcervical arterial ligation on the severity of postoperative hemorrhage after transoral robotic surgery. Head Neck. 2017 Aug;39(8):1510-1515. doi: 10.1002/hed.24677. Epub 2017 Jun 1. PMID 28570011
- [Background] Hay A, Migliacci J, Karassawa Zanoni D, Boyle JO, Singh B, Wong RJ, Patel SG, Ganly I. Haemorrhage following transoral robotic surgery. Clin Otolaryngol. 2018 Apr;43(2):638-644. doi: 10.1111/coa.13041. Epub 2017 Dec 26. PMID 29194991
- [Background] Gleysteen J, Troob S, Light T, Brickman D, Clayburgh D, Andersen P, Gross N. The impact of prophylactic external carotid artery ligation on postoperative bleeding after transoral robotic surgery (TORS) for oropharyngeal squamous cell carcinoma. Oral Oncol. 2017 Jul;70:1-6. doi: 10.1016/j.oraloncology.2017.04.014. Epub 2017 May 9. PMID 28622885
- [Background] Mehanna H, Evans M, Beasley M, Chatterjee S, Dilkes M, Homer J, O'Hara J, Robinson M, Shaw R, Sloan P. Oropharyngeal cancer: United Kingdom National Multidisciplinary Guidelines. J Laryngol Otol. 2016 May;130(S2):S90-S96. doi: 10.1017/S0022215116000505. PMID 27841123
- [Background] Robinson AE, McAuliffe W, Phillips TJ, Phatouros CC, Singh TP. Embolization for the treatment of intractable epistaxis: 12 month outcomes in a two centre case series. Br J Radiol. 2017 Dec;90(1080):20170472. doi: 10.1259/bjr.20170472. Epub 2017 Oct 26. PMID 28972795
- [Background] Gemmete JJ, Ansari SA, McHugh J, Gandhi D. Embolization of vascular tumors of the head and neck. Neuroimaging Clin N Am. 2009 May;19(2):181-98, Table of Contents. doi: 10.1016/j.nic.2009.01.008. PMID 19442905
- [Background] Kai Y, Hamada J, Morioka M, Yano S, Todaka T, Ushio Y. Appropriate interval between embolization and surgery in patients with meningioma. AJNR Am J Neuroradiol. 2002 Jan;23(1):139-42. PMID 11827886
- [Background] Chun JY, McDermott MW, Lamborn KR, Wilson CB, Higashida R, Berger MS. Delayed surgical resection reduces intraoperative blood loss for embolized meningiomas. Neurosurgery. 2002 Jun;50(6):1231-5; discussion 1235-7. doi: 10.1097/00006123-200206000-00010. PMID 12015840
- [Background] Schrock A, Jakob M, Strach K, Pump B, Gerstner AO, Wilhelm K, Urbach H, Bootz F, Greschus S. Transarterial endovascular treatment in the management of life-threatening intra- and postoperative haemorrhages after otorhinolaryngological surgery. Eur Arch Otorhinolaryngol. 2012 Jun;269(6):1677-83. doi: 10.1007/s00405-011-1823-4. Epub 2011 Nov 12. PMID 22081095
- [Background] Wong DJY, Donaldson C, Lai LT, Coleman A, Giddings C, Slater LA, Chandra RV. Safety and effectiveness of endovascular embolization or stent-graft reconstruction for treatment of acute carotid blowout syndrome in patients with head and neck cancer: Case series and systematic review of observational studies. Head Neck. 2018 Apr;40(4):846-854. doi: 10.1002/hed.25018. Epub 2017 Nov 20. PMID 29155470
- [Background] Cohen JE, Moscovici S, Gomori JM, Eliashar R, Weinberger J, Itshayek E. Selective endovascular embolization for refractory idiopathic epistaxis is a safe and effective therapeutic option: technique, complications, and outcomes. J Clin Neurosci. 2012 May;19(5):687-90. doi: 10.1016/j.jocn.2011.08.019. Epub 2012 Feb 23. PMID 22364712
- [Background] de Bonnecaze G, Gallois Y, Bonneville F, Vergez S, Chaput B, Serrano E. Transnasal Endoscopic Sphenopalatine Artery Ligation Compared With Embolization for Intractable Epistaxis: A Long-term Analysis. Am J Rhinol Allergy. 2018 May;32(3):188-193. doi: 10.1177/1945892418768584. Epub 2018 Apr 20. PMID 29676168